CLINICAL TRIAL: NCT03702712
Title: Acute Effects of Aerobic Exercise and Relaxation on Fatigue and Executive Function in Breast Cancer Survivors
Brief Title: Responsiveness to Acute Changes in Exercise and Relaxation (RACER) Trial
Acronym: RACER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Sean Mullen, Associate Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16381
Record Dates: First submitted 2018-10-03; First posted 2018-10-11 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer
Keywords: Survivorship; Fatigue; Relax; Cognition; Exercise
MeSH Terms: conditions — Breast Neoplasms; Fatigue; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic Exercise Only (Active Comparator): Participants in the Aerobic Exercise Only arm will engage in three separate 20-minute sessions comprised of a 5-minute, resistance-free warm-up, and 15 minutes of moderate stationary aerobic cycling on a Cybex bike #525C (50-70% age-predicted heart rate max). Each session will be followed by 20 minutes of uninterrupted quiet rest. The bike will provide feedback including speed, rotations per minute, and time.
  Interventions: Behavioral: Aerobic Exercise Only
- Relaxation Only (Active Comparator): Participants in the Relaxation Only arm will complete three separate 20-minute sessions of relaxation using a commercial wearable neurofeedback (headband) device. The device's accompanying software (connected to the headband through Bluetooth) encourages breathing strategies in response to recorded brain wave activity. Real time auditory feedback includes sounds of calm (soft) or loud winds in response to detected brain activity. A visual report of affective states and the user's brain activity is given (alpha and beta waves). Participants will also be asked to take part in 20 minutes of uninterrupted quiet rest in order to match the time of the aerobic only condition.
  Interventions: Behavioral: Relaxation Only
- Aerobic Exercise and Relaxation (Experimental): Participants in the Aerobic Exercise and Relaxation arm will complete the three separate 20-minute aerobic exercise sessions (identical to the aerobic exercise only condition) followed by the same 20-minute neurofeedback-guided mindfulness training (identical to the relaxation only condition).
  Interventions: Behavioral: Aerobic Exercise and Relaxation

INTERVENTIONS:
Behavioral: Aerobic Exercise and Relaxation — This intervention will combine 20 minutes of moderate aerobic exercise followed by 20 minutes of mindfulness training.
  Arms: Aerobic Exercise and Relaxation
Behavioral: Aerobic Exercise Only — This intervention will combine 20 minutes of moderate aerobic exercise followed by 20 minutes of quiet rest.
  Arms: Aerobic Exercise Only
Behavioral: Relaxation Only — This intervention will combine 20 minutes of mindfulness-based relaxation training followed by 20 minutes of quiet rest.
  Arms: Relaxation Only

SUMMARY:
The purpose of this acute study is to compare the combined effects of aerobic exercise and relaxation training on fatigue and its related cognitive components, among breast cancer survivors. Participants will complete three sessions over a seven-day period in a laboratory setting.

DETAILED DESCRIPTION:
It is hypothesized that the combination of aerobic exercise and relaxation training could have additive effects on fatigue and related cognitive outcomes. Therefore, this study is designed to test the effects of exercise plus relaxation relative to aerobic exercise alone and relaxation training alone, over the course of three sessions within a seven day period. Participants will complete baseline and post-testing before and after the week of training, as well as pre- and post-testing at each session.

Participants will be randomized to one of three conditions:

1. Aerobic Exercise Only Condition (AERO) Participants randomized to the AERO condition will engage in three separate 20-minute sessions comprised of a 5-minute, resistance-free warm-up, and 15 minutes of moderate aerobic cycling on a stationary bike (50-70% age-predicted heart rate max). Each AERO session will end with a 20-minute quiet rest period.
2. Relaxation Only Condition (RELAX) Participants in the RELAX condition will complete three separate 20-minute sessions of relaxation training using a commercial neurofeedback device (headset & smartphone app). Each RELAX session will end with a 20-minute quiet rest period.
3. Aerobic Exercise and Relaxation Training - Intervention Condition (COMBINED) Participants randomized to the COMBINED condition will complete three separate sessions comprised of 20 minutes of AERO exercise followed by 20 minutes of RELAX training.

All participants, regardless of condition will complete brief questionnaires assessing in-the-moment fatigue and affect, before and after each randomly assigned activity session. A larger survey and battery of cognitive tests will be completed at the beginning of the first appointment and at the conclusion of the third appointment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* previously diagnosed with breast cancer (ductal carcinoma in situ or stages I-IV)
* completed at least one cycle of chemotherapy treatment within the last 5 years
* must have reliable access to the internet
* must report at least one complaint concerning physical function, fatigue, memory, planning, thinking, negative mood, depressive symptoms, or anxiety
* must be capable of engaging in sustained stationary cycling at a moderate intensity

Exclusion Criteria:

* deaf in both ears
* unable to comfortably wear a pair of ear-bud headphones
* color-blind or do not have vision of at least 20/40 with the aid of contacts or glasses
* history or diagnosis of epilepsy

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only individuals who identify as female who have survived breast cancer (in situ, stages I-IV) will be recruited.
Enrollment: 40 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Piper Fatigue Scale | This will be assessed on day 1 (baseline), day 2 and day 3 (post-testing), both before and after randomized activities.
  The Piper Fatigue Scale requires respondents to select their answers according to a "0" (most positive or desirable response) to "10" (most negative, fatigue is having a strong impact) scale. A total fatigue score is calculated by summing each of the 12 responses and dividing by 12. Accordingly, a total fatigue change score of 0 corresponds to no fatigue, a score of 1-3 is labeled as mild, 4-6 is labeled as moderate, and 7-10 is labeled as severe. The total scores from each of the three days will be used to calculate an overall fatigue score, which will be used to assess group level differences across averages. Our operational definition of overall fatigue in this outcome is the average score across each group.

SECONDARY OUTCOMES:
Perceived Mental Fatigue | The PMFQ will be assessed on day 1 (baseline), day 2, and day 3 (post-testing).
  The Perceived Mental Fatigue Questionnaire (PMFQ) is a novel inventory using 7-item Likert scale ( e.g., "My thinking requires effort," 1 = Not at all to 5 = Very true). Participants are asked to reflect on their current level of mental fatigue. The 7 items from PMFQ are summed together to create a composite fatigue value. The total scores from each of the three days will be used to calculate an overall fatigue score, which will be used to assess group level differences across averages. Our operational definition of overall fatigue in this outcome is the average score across each group.
Energy subscale of AD ACL-SAI | This will be assessed following randomized activities on Day 1 (baseline), Day 2, and Day 3 (post-testing).
  The AD ACL-SAI asks respondents to select how they relate to a specific adjective in the moment by choosing between 4 answer options (1=not at all, 2=moderately so, 3=somewhat, and 4=very much so). Each of the 5 items in the Energy subscale are summed together to create an overall Energy fatigue score.The total scores from each of the three days will be used to calculate an overall energy score, which will be used to assess group level differences across averages. Our operational definition of overall energy in this outcome is the average score across each group.
Tiredness subscale of AD ACL-SAI | This will be assessed following randomized activities on Day 1 (baseline), Day 2, and Day 3 (post-testing).
  The AD ACL-SAI asks respondents to select how they relate to a specific adjective in the moment by choosing between 4 answer options (1=not at all, 2=moderately so, 3=somewhat, and 4=very much so). Each of the 5 items in the Tiredness subscale are summed together to create an overall Tiredness fatigue score. This will be used to calculate a change score. The total scores from each of the three days will be used to calculate an overall tiredness score, which will be used to assess group level differences across averages. Our operational definition of overall tiredness in this outcome is the average score across each group.
Attention- Assessed by Flanker Inhibitory Control and Attention task from the NIH toolbox | This will be assessed prior to randomized activities on day 1 (baseline), and day 3 (post-testing)
  In the Flanker task participants focus on a given stimulus while inhibiting attention to stimuli flanking it. Participants see a row of 5 arrows and choose the button that matches the direction the middle arrow is pointing. This test yields a standardized accuracy and processing speed change score.
Working Memory- Assessed by Picture Sequence task from the NIH toolbox | This will be assessed prior to randomized activities on day 1 (baseline), and day 3 (post-testing)
  The Picture Sequence tasks asks participants to remember a specific order of events as demonstrated by the task itself on a screen. At the conclusion of the demonstration, the events are scrambled and the participants are instructed to place them back in the correct order. This task yields a standardized accuracy change score.
Cognitive Flexibility and Attention- Assessed by Dimensional Change Card Sort Task from the NIH toolbox | This will be assessed prior to randomized activities on day 1 (baseline), and day 3 (post-testing)
  In the Dimensional Change Card Sort Task, participants are asked to match a series of bivalent test pictures (e.g., yellow balls and blue trucks) to the target pictures, first according to one dimension (e.g., color) and then, after a number of trials, according to the other dimension (e.g., shape). The ensuing "switch" trials are also employed, in which the participant is required to change the dimension being matched. For example, after 4 straight trials matching on shape, the participant may be asked to match on color on the next trial and then go back to shape, thus requiring the cognitive flexibility to quickly choose the correct stimulus. The NIH toolbox automatically calculates an overall raw score, which takes into account both accuracy and reaction time, used to create a change score.
Program Evaluation - Perceived Usefulness | This will be assessed on day 3.
  All participants will complete an adapted version of Davis (1989) and Davis et al., (1989) perceived usefulness questionnaire (e.g., "Using the technology-delivered relaxation training program improved my thinking"). These 5 items will be measured using a 7-point Likert scale (1 = Strongly disagree, 4 = Neutral, 7 = Strongly agree) and will assess attitudes towards the technology-delivered relaxation-training program. The 5 item's responses will be averaged and then used for a total perceived usefulness score.
Program Evaluation - Perceived Ease of Use | This will be assessed on day 3.
  All participants will complete an adapted version of Davis (1989) and Davis et al., (1989) perceived ease of use questionnaire (e.g., "I found the technology-delivered relaxation training program to be easy to use"). These 5 items will be measured using a 7-point Likert scale (1 = Strongly disagree, 4 = Neutral, 7 = Strongly agree) and will assess attitudes towards the technology-delivered relaxation-training program. The 5 item's responses will be averaged and then used for a total perceived usefulness score.
Program Evaluation - Enjoyment | This will be assessed on day 3.
  An evaluation of participants' enjoyment of the trial will also be included. Five questions (e.g., I enjoyed using the mindfulness training device) using a 7-point Likert scale (1 = Not at all, 4 = Neutral, 7 = Completely) will be administered. The 5 item's responses will be averaged and then used for a total perceived usefulness score.
Program Evaluation - Satisfaction | This will be assessed on day 3.
  An evaluation of participants' satisfaction with components of the trial will also be included. Five questions (e.g., I am satisfied with the outcomes experienced following mindfulness training) using a 7-point Likert scale (1 = Not at all, 4 = Neutral, 7 = Completely) will be administered. The 5 item's responses will be averaged and then used for a total perceived usefulness score.
Program Evaluation - Open Ended | This will be assessed on day 3.- focusing on thoughts of the program over the three appointment days, in a 1-week period.
  An open ended evaluation of participants' experience with the trial will also be included. This qualitative question will ask participants to expand upon their overall likes and dislikes, recommendations, and modifications will be included. Open ended responses will be used to design and apply future interventions in this area.

CONTACTS AND LOCATIONS:
Overall Officials: Sean P Mullen, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- University of Illinois at Urbana-Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be made available for all primary and secondary outcome measures. Included documentation will be comprised of study protocol, statistical analyses protocols, informed consent documentation, and layperson research procedures. Additionally information will be made available upon request. Data access requests will be reviewed by the primary investigators. Requestors will be required to sign a Data Access Agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Although this is not an NIH funded study, we will update these records within 1 year of data collection completion per NIH guidelines.
Access Criteria: Data will be accessible on an open site (e.g., Open Science Framework https://osf/io/) with a request to interested parties to engage with the investigative team about any publication of these data in an effort to avoid redundancy. Appropriate authorship crediting investigators involved in the parent study conceptualization, and any consultation regarding data interpretation should be sought by any researchers interested in publishing these data.

REFERENCES:
- [Derived] Cohen J, Rogers WA, Petruzzello S, Trinh L, Mullen SP. Acute effects of aerobic exercise and relaxation training on fatigue in breast cancer survivors: A feasibility trial. Psychooncology. 2021 Feb;30(2):252-259. doi: 10.1002/pon.5561. Epub 2020 Oct 14. PMID 33010183
- See also: Exercise, Technology, and Cognition Laboratory — http://exercisetechlab.com